CLINICAL TRIAL: NCT02556164
Title: Objective Assessment of Electro-acupuncture Efficacy for Gait and Balance in Patients With Parkinson's Disease
Brief Title: Electro-acupuncture for Gait and Balance in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Hong Lei, Associate Professor of Clinical Neurology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UArizona
Record Dates: First submitted 2015-09-08; First posted 2015-09-22 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Parkinson's Disease
Keywords: Electroacupuncture; Body Worn Sensor; Gait; Balance
MeSH Terms: conditions — Parkinson Disease | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real EA (Experimental): Real EA as intervention is performed at the selected standard acupuncture points and "De-qi" is achieved with needle manipulation before electric stimulation is delivered.
  Interventions: Procedure: Electroacupuncture; Other: Body-worn sensor technology
- Sham EA (Sham Comparator): Sham EA as intervention is performed for the control group at non-acupuncture points without needle manipulation. The electric stimulation in sham acupuncture was performed in a similar fashion to the real EA.
  Interventions: Procedure: Electroacupuncture; Other: Body-worn sensor technology

INTERVENTIONS:
Procedure: Electroacupuncture — Acupuncture is an alternative medicine methodology that treats patient by various techniques including inserting small, thin needles at specific points of body. Electroacupuncture (EA), like the name implies, combines classical acupuncture and low electric current running through the needles, which are often used to enhance a treatment.
Other: Body-worn sensor technology — Three-dimensional acceleration and angular velocity of shanks, thighs and the trunk were measured using wearable sensors each included a triaxial accelerometer and a triaxial gyroscope (LEGSys™ and BalanSens™ - BioSensics, Boston, MA)

SUMMARY:
Gait and balance disorders, key contributors to fall and poor quality of life, represent a major therapeutic challenge in Parkinson's disease (PD). Despite the widespread use of acupuncture in recent years in PD, its efficacy remains unclear, largely due to methodological flaws and lack of high quality studies using objective outcome measures. In a patient and assessor-blind pilot study, investigators objectively assess the efficacy of electroacupuncture (EA) for gait and balance disorders using body-worn sensor technology in patients with PD.

DETAILED DESCRIPTION:
In this study, investigators employee objective innovative body-worn sensor technologies to assess potential mobility-associated outcomes of PD. Investigators compare acute changes in gait and balance that occurred after repeated administration of two interventions: A specific real EA and a sham EA. The design of the experiments uses a control that accounts for both placebo and possible some active components of a generalized needle-insertion-based procedure. By using a sham control, the investigators were able to more fully test whether the specific EA intervention could lead to changes in objective gait and balance parameters, or subjective self-reported improvements that are beyond placebo induced effects and the natural course of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling men or women ages 55 years or older with diagnosis of PD;
2. patients who have the ability to walk 20meters without walking assistance; and
3. patients who are stable without anti-PD medication(s) change for at least 1 month. The PD diagnosis was made by movement disorder specialists based on the UK Brain Bank criteria and supported by DaTscan (Ioflupane I 123 injection) when possible.

Exclusion Criteria:

1. patients who have received previous acupuncture;
2. patients who have had DBS;
3. patients with any clinically significant medical condition, psychiatric condition, drug or alcohol abuse, or laboratory abnormality that would, in the judgment of the investigators, interfere with the ability to participate in the study; and
4. patients with non-PD related gait disorders.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2016-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change of gait speed by objective measurement | 3 weeks
  Participant performs two tests of normal gait (> 25 steps) under single task and dual task conditions. Gait speed (m/s) is assessed using body-worn sensor technology.

SECONDARY OUTCOMES:
Change of postural balance (COG) by objective measurement | 3 weeks
  Each participant performs 30-second trials of balance assessment with eyes open or closed. Center of gravity (COG, cm) is assessed using body-worn sensor technology.
Change of stride length by objective measurement | 3 weeks
  Participant performs two tests of normal gait (> 25 steps) under single task and dual task conditions. Stride length (m) is assessed using body-worn sensor technology.
Change of postural balance (Ankle/hip sway) by objective measurement | 3 weeks
  Each participant performs 30-second trials of balance assessment with eyes open or closed. Ankle sway (deg2), Hip sway (deg2), Ankle/hip sway is assessed using body-worn sensor technology.
Change of Unified Parkinson's Disease Rating Scale | 3 weeks
  Unified Parkinson's disease rating scale (UPDRS) is utilized. Parts I: to assess mentation, behavior and mood (0-16); Part II: to assess activities of daily living ( 0-52); Part III to motor assessment (0-104)
Change of SF-12 health survey | 3 weeks
  SF-12 health survey (MCS, PCS)
Change of Short Falls Efficacy Scale-International | 3 weeks
  (Short FES-I, 7-28)
Change of the visual analog scale | 3 weeks
  the visual analog scale (VAS, 0-10) for pain,
Potential adverse events related to acupuncture | Baseline, 1 week, 2 week and 3 weeks.
  measured by Adverse Events Report Related to Acupuncture

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Najafi, PhD, Principal Investigator — University of Arizona

REFERENCES:
- [Derived] Lei H, Toosizadeh N, Schwenk M, Sherman S, Karp S, Sternberg E, Najafi B. A Pilot Clinical Trial to Objectively Assess the Efficacy of Electroacupuncture on Gait in Patients with Parkinson's Disease Using Body Worn Sensors. PLoS One. 2016 May 26;11(5):e0155613. doi: 10.1371/journal.pone.0155613. eCollection 2016. PMID 27227460